CLINICAL TRIAL: NCT03661879
Title: A Randomised, Double-blinded, Multiple-dose Trial Investigating Safety, Tolerability and Pharmacokinetics of NNC9204-1706 in Subjects Being Overweight or With Obesity
Brief Title: Research Study of a New Medicine (NNC9204-1706) in People With Overweight or Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9423-4393; U1111-1208-7677 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-09-05; First posted 2018-09-07 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-10

CONDITIONS: Metabolism and Nutrition Disorder; Obesity
MeSH Terms: conditions — Nutrition Disorders; Obesity

STUDY DESIGN:
Intervention Model Description: Five (5) cohorts are planned. In each cohort, subjects will be randomised in a 3:1 manner to receive either: 1) NNC9204-1706: 9 subjects or 2) Placebo (NNC9204-1706): 3 subjects
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC9204-1706 (Experimental): Participants will receive NNC9204-1706 for 10 weeks. There will be a 2-week follow-up period after the treatment period.
  Interventions: Drug: NNC9204-1706
- Placebo (NNC9204-1706) (Placebo Comparator): Participants will receive placebo (NNC9204-1706) for 10 weeks. There will be a 2-week follow-up period after the treatment period.
  Interventions: Drug: Placebo (NNC9204-1706)

INTERVENTIONS:
Drug: NNC9204-1706 — Participants will receive NNC9204-1706 subcutaneous (s.c., under the skin) injection(s) once daily (OD) for 10 weeks. They will either receive the same dose throughout the trial, or the dose will be escalated over a period of 1-3 weeks and continued for at least 7 weeks at the same dose.
  Arms: NNC9204-1706
Drug: Placebo (NNC9204-1706) — Participants will receive matching placebo (NNC9204-1706) s.c., injection(s) OD for 10 weeks.
  Arms: Placebo (NNC9204-1706)

SUMMARY:
The study is testing a new medicine for weight control in people with overweight or obesity. The aim of the study is to find out how safe the study medicine is and how it works in the body. Participants will either get NNC9204-1706 (the new study medicine) or placebo (a dummy medicine) - which treatment participants get is decided by chance. NNC9204-1706 is a new medicine which cannot be prescribed by doctors. Participants will get an injection under the skin of participants' stomach each morning for 10 weeks. A medical tool called NovoPen®4 will be used for the injection. Participants must change the part of the pen including the medicine (the cartridge) each day. The study will last for about 16 weeks. Participants will have at least 17 clinic visits and 10 phone calls with the study doctor. At certain times during the study, participants will have blood drawn and 3 different kinds of heart tests (electrocardiograms). Study doctor will ask participants to answer mental health surveys.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 25.0 and 39.9 kg/m^2 (both inclusive) at screening. Overweight should be due to excess adipose tissue, as judged by the investigator.

Exclusion Criteria:

* Female subject who is of childbearing potential (pre-menopausal and not surgically sterilised) and is sexually active with male partner(s) who are not surgically sterilised (vasectomy) or who is not using highly effective contraceptive methods (Pearl Index less than 1%) combined with a highly effective method of contraception for their male partner(s) (e.g. condom with spermicide), or are pregnant, breast-feeding or intend to become pregnant.
* Male subject who is not surgically sterilised (vasectomy) and is sexually active with female partner(s) and who is not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their nonpregnant female partner(s) (Pearl Index less than 1%), and/or intend to donate sperm in the period from screening until 90 days following administration of the investigational medical product.
* Any disorder which in the investigator's opinion might jeopardise subject's safety, evaluation of results, or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-09-12 (Actual); Primary Completion 2019-09-05 (Actual); Study Completion 2019-10-09 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | Days 1-84
  Count of adverse events.

SECONDARY OUTCOMES:
Change in time-profile (msec) in individual corrected QT interval (ΔQTcI) | Day 1, Day 84
  Measured in msec.
AUC0-24h,SS (h*nmol/L); the area under the NNC9204-1706 plasma concentration-time curve from time 0 to 24 hours at steady state | Days 1-84
  Measured in h*nmol/L.
Cmax,SS (nmol/L); the maximum plasma concentration of NNC9204-1706 at steady state | Days 1-84
  Measured in nmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results

REFERENCES:
- [Derived] Skovgaard D, Haahr PM, Lester R, Clark K, Paglialunga S, Finer N, Friedrichsen MH, Hjerpsted JB, Engelmann MDM. Prevalence of Baseline Cardiac Arrhythmias in Participants with Overweight or Obesity in Phase 1 Clinical Trials: Analysis of 24-Hour Holter Electrocardiogram Recordings. J Clin Pharmacol. 2023 May;63(5):539-543. doi: 10.1002/jcph.2193. Epub 2023 Jan 20. PMID 36524539